CLINICAL TRIAL: NCT01387412
Title: The Role of Genital Warts in HIV Acquisition Among MSM in Peru"
Brief Title: The Role of Genital Warts in HIV Acquisition in Peru
Acronym: VIVA
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Espacio Comun (Unknown); Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Brandon Brown, Faculty, University of California, Los Angeles
Other Study IDs: Merck IISP 39619
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Anogenital Warts; HIV
Keywords: genital warts; HIV; MSM; Peru; HPV
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, lesion biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Genital warts: Those with and without ano-genital warts

SUMMARY:
The primary objective of this study is to determine the role of genital warts (GW) on Human Immunodeficiency Virus (HIV) acquisition among men who have sex with men (MSM) in Peru. The secondary objectives are to determine Human Papillomavirus (HPV) prevalence in HIV positive MSM in Peru, risk factors associated with GW, and the knowledge of HPV and HIV among MSM.

DETAILED DESCRIPTION:
Persons with Human Immunodeficiency Virus (HIV) infection are at higher risk of becoming infected with the Human Papillomavirus (HPV) compared to those who are HIV negative. The contrary is also true: individuals infected with HPV may be more likely to acquire HIV; however, the role of the clinical manifestation of HPV - genital warts (GW) - on HIV acquisition is currently unknown. Few studies have shown that GW are independently associated with HIV acquisition.

The primary objective of this study is to determine the role of GW on HIV acquisition among MSM in Peru. The secondary objectives are to determine HPV prevalence in HIV positive MSM in Peru, risk factors associated with GW, and the knowledge of HPV and HIV among MSM. The specific aims of this study are:

1. To estimate HIV incidence in Peruvian MSM by GW status.
2. To determine the prevalence of HIV among Peruvian MSM by GW status.
3. To determine the type-specific prevalence of anal HPV infection in HIV positive Peruvian MSM. Linear array testing will estimate prevalence of 37 HPV types including carcinogenic (16,18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66) and non-carcinogenic types (6, 11, 26, 40, 42, 53, 54, 61, 62, 64, 67, 68, 69, 70, 72, 73, 81, 82, 82var, 83, 84, and 89) as defined at the 2005 meeting of the International Agency for Research on Cancer.
4. To identify risk factors associated with genital warts (penile, anal, and both) among Peruvian MSM.
5. To assess the knowledge of Peruvian MSM of the role of HPV in HIV infection.

The study will be conducted in the Gay Men's Community Health Center, Epicentro, the only center in Lima that specifically caters to men who have sex with men and sees a high burden of genital warts in their patient population. The study includes a population of 600 MSM (300 with recent or current genital warts). Baseline HIV serostatus will be done by rapid testing, and follow-up for HIV incidence will be done every 6 months over a two year time period. We will determine HPV status in HIV-positive participants and refer them for free highly active antiretroviral therapy (HAART) treatment. We will examine participants for GW presence and collect information on history of GW. A survey will be administered at each visit which examines changes in risk behaviors over time.

This novel study proposes to both measure the prevalence of GW in MSM presenting at a community clinic environment and prospectively measure HIV incidence in men with GW and those without GW. It will be the first study of its kind that we are aware of using HIV infection as an endpoint in men with and without GW and will help to better understand the relationship between genital warts and HIV infection among MSM in Peru.

ELIGIBILITY:
Inclusion Criteria:

* Anatomical males 18-40 years of age,
* Self-reported anal sex with another man within 12 months prior to enrollment,
* Willing to provide informed consent for the collection of demographic and sexual behavior data, as well as blood for HIV and Syphilis testing, swabs of anal mucosa for HPV testing and urine for Chlamydia testing,
* Resident of metropolitan Lima.

Exclusion Criteria:

* Prior participation in an HPV vaccine clinical trial,
* Prior participation in an HIV vaccine clinical trial,
* Presence of a known immunodeficiency that increases risk of acquiring HIV.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
HIV incidence | 2 years
  new cases of HIV in our cohort in either the group with or without genital warts

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Brown, PhD, Principal Investigator — University of California, Los Angeles; Jerome Galea, MSW, Study Director — Espacio Comun
Locations (1):
- Espacio Comun, Barranco, Lima region, Peru

REFERENCES:
- [Background] Smith JS, Moses S, Hudgens MG, Parker CB, Agot K, Maclean I, Ndinya-Achola JO, Snijders PJ, Meijer CJ, Bailey RC. Increased risk of HIV acquisition among Kenyan men with human papillomavirus infection. J Infect Dis. 2010 Jun 1;201(11):1677-85. doi: 10.1086/652408. PMID 20415595
- [Background] Jin F, Prestage GP, Imrie J, Kippax SC, Donovan B, Templeton DJ, Cunningham A, Mindel A, Cunningham PH, Kaldor JM, Grulich AE. Anal sexually transmitted infections and risk of HIV infection in homosexual men. J Acquir Immune Defic Syndr. 2010 Jan;53(1):144-9. doi: 10.1097/QAI.0b013e3181b48f33. PMID 19734801
- [Background] Caceres CF, Mendoza W. Monitoring trends in sexual behaviour and HIV/STIs in Peru: are available data sufficient? Sex Transm Infect. 2004 Dec;80 Suppl 2(Suppl 2):ii80-4. doi: 10.1136/sti.2004.012021. PMID 15572646
- [Background] Bautista CT, Sanchez JL, Montano SM, Laguna-Torres VA, Lama JR, Sanchez JL, Kusunoki L, Manrique H, Acosta J, Montoya O, Tambare AM, Avila MM, Vinoles J, Aguayo N, Olson JG, Carr JK. Seroprevalence of and risk factors for HIV-1 infection among South American men who have sex with men. Sex Transm Infect. 2004 Dec;80(6):498-504. doi: 10.1136/sti.2004.013094. PMID 15572623
- [Background] Clark JL, Segura ER, Montano SM, Leon SR, Kochel T, Salvatierra HJ, Alcantara J, Caceres CF, Coates TJ, Klausner JD. Routine laboratory screening for acute and recent HIV infection in Lima, Peru. Sex Transm Infect. 2010 Dec;86(7):545-7. doi: 10.1136/sti.2010.042697. PMID 21113069
- [Background] Goldstone S, Palefsky JM, Giuliano AR, Moreira ED Jr, Aranda C, Jessen H, Hillman RJ, Ferris DG, Coutlee F, Liaw KL, Marshall JB, Zhang X, Vuocolo S, Barr E, Haupt RM, Guris D, Garner EI. Prevalence of and risk factors for human papillomavirus (HPV) infection among HIV-seronegative men who have sex with men. J Infect Dis. 2011 Jan 1;203(1):66-74. doi: 10.1093/infdis/jiq016. PMID 21148498
- [Background] Li AH, Phanuphak N, Sahasrabuddhe VV, Chaithongwongwatthana S, Vermund SH, Jenkins CA, Shepherd BE, Teeratakulpisarn N, van der Lugt J, Avihingsanon A, Ruxrungtham K, Shikuma C, Phanuphak P, Ananworanich J. Anal squamous intraepithelial lesions among HIV positive and HIV negative men who have sex with men in Thailand. Sex Transm Infect. 2009 Dec;85(7):503-7. doi: 10.1136/sti.2009.036707. Epub 2009 Jun 11. PMID 19525263
- [Background] Cohen MS. Sexually transmitted diseases enhance HIV transmission: no longer a hypothesis. Lancet. 1998;351 Suppl 3:5-7. doi: 10.1016/s0140-6736(98)90002-2. No abstract available. PMID 9652712
- [Background] Fleming DT, Wasserheit JN. From epidemiological synergy to public health policy and practice: the contribution of other sexually transmitted diseases to sexual transmission of HIV infection. Sex Transm Infect. 1999 Feb;75(1):3-17. doi: 10.1136/sti.75.1.3. PMID 10448335
- [Background] Grosskurth H, Mosha F, Todd J, Mwijarubi E, Klokke A, Senkoro K, Mayaud P, Changalucha J, Nicoll A, ka-Gina G, et al. Impact of improved treatment of sexually transmitted diseases on HIV infection in rural Tanzania: randomised controlled trial. Lancet. 1995 Aug 26;346(8974):530-6. doi: 10.1016/s0140-6736(95)91380-7. PMID 7658778
- [Derived] Flores JA, Brown B, Leon SR, Sanchez H, Galea JT. Individual-level characteristics associated with oral HIV test acceptability among Peruvian men who have sex with men and transgender women: a cross-sectional study. Sex Transm Infect. 2018 Nov;94(7):528-533. doi: 10.1136/sextrans-2017-053388. Epub 2018 Mar 24. PMID 29574465
- [Derived] Galea JT, Leon SR, Peinado J, Calvo G, Zamora J, Sanchez H, Brown BJ. HPV knowledge, burden and genital wart location among heterosexually identified versus homosexually identified men who have sex with men in Lima, Peru: cross-sectional results from a cohort study. BMJ Open. 2017 Oct 24;7(10):e017338. doi: 10.1136/bmjopen-2017-017338. PMID 29070638
- [Derived] Brown B, Davtyan M, Leon SR, Sanchez H, Calvo G, Klausner JD, Galea J. A prospective cohort study characterising the role of anogenital warts in HIV acquisition among men who have sex with men: a study protocol. BMJ Open. 2014 Sep 16;4(9):e005687. doi: 10.1136/bmjopen-2014-005687. PMID 25227629